CLINICAL TRIAL: NCT04956887
Title: Cognitive Training in Survivors of Covid-19: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, James C. Jackson, Research Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 210121
Record Dates: First submitted 2021-07-07; First posted 2021-07-09 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Covid19; Cognitive Impairment
MeSH Terms: conditions — COVID-19; Cognitive Dysfunction | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: After the patient or authorized surrogate provides informed consent, the cognitive training and rehabilitation intervention versus usual care will be randomly assigned at a 1:1 allocation ratio. Computerized randomization will occur after informed consent has been obtained using a permuted-block randomization scheme with varying block size. We will use adequate allocation concealment using a computer-generated, permuted-block randomization scheme with varying block size. The block size and randomization list will only be known to the independent biostatistician creating the randomization list and will not be shared with trial investigators or any other study personnel, as this information could make it easier to correctly guess the next treatment allocation. This list will be directly uploaded into REDCap's randomization module.16
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The study intervention, AKL-T01 (Akili Interactive), is a digital, app-based intervention designed to target and improve cognition through an engaging video game-based software experience delivered on an iPad.
  Interventions: Behavioral: AKL-T01
- Placebo (Placebo Comparator): Patients assigned to the control group will receive no intervention, as is typical for those with Covid-19 with respect to cognitive functioning.
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: AKL-T01 — The study intervention, AKL-T01 (Akili Interactive), is a digital, app-based intervention designed to target and improve cognition through an engaging video game-based software experience delivered on an iPad.
  Arms: Intervention
Other: Control Group — Patients assigned to the control group will receive no intervention, as is typical for those with Covid-19 with respect to cognitive functioning
  Arms: Placebo

SUMMARY:
Preliminary evidence suggests that cognitive impairment is a common outcome experienced by individuals surviving Covid-19 (1-5). Cognitive impairment following Covid-19 which leads to critical illness is not surprising and perhaps even expected. However, significant cognitive deficits appear to be common even among individuals testing positive for Covid-19 who were never hospitalized. Questions exist regarding the mechanisms of the aforementioned cognitive impairment. The association between COVID-19 and brain dysfunction is not surprising since SARS-CoV has been found in the brain and because Coronaviridaes (CoVs) have been associated with central nervous system (CNS) diseases such as acute viral encephalopathy, acute disseminated encephalomyelitis, and multiple sclerosis (6-11).The possible brain entry routes for CoVs include either direct intranasal access to the brain via olfactory nerves or indirect access by crossing the blood-brain barrier (BBB) via hematogenous or lymphatic spread (9).

DETAILED DESCRIPTION:
As the Investigators have described, a frequent and particularly disabling consequence of Covid-19 may be in the cognitive arena, with deleterious implications for employment, quality of life, and other dimensions of functioning. As such, efforts to develop interventions aimed at improving neuropsychological outcomes are important and a key feature of an overarching public health strategy. One potential intervention of interest is cognitive training, which has been employed with increasing success with wide-ranging populations, though only minimally with survivors of critical illness and not with Covid-19 patients at all. Cognitive training, particularly the kind that relies on what are known as digital interventions (programs which, functionally, look like video games) is particularly appropriate in the pandemic climate, as it can be done entirely in a virtual contactless fashion, thus decreasing the risk of infection. The Investigators propose a pilot study in 100 cognitively impaired community dwelling patients who tested positive for Covid-19 and are participants in an existing study/ongoing study of household transmission of Covid-19 (the SARS-Co-V-2 Household Transmission Study, with the following specific aim and hypotheses:

Study Aim: To evaluate the feasibility of conducting a randomized trial evaluating the effectiveness of a digital app-based intervention (AKL-T01) to improve 4-week cognition (post-intervention) in cognitively impaired survivors of Covid-19.

Hypothesis 1: A trial evaluating AKL-T01 for improving long-term cognition in community dwelling and cognitively abnormal COVID-19 patients will be feasible, as denoted by achieving each of the following in this pilot trial: (a) recruitment and successful protocol completion of up to 100 patients; (b) successful completion of 4-week cognitive assessments by >80% of survivors; and (c) the primary cognitive outcome (a composite score on CNS Vital Signs) numerically favoring the intervention group with the one-tailed upper 80% confidence interval of the difference in a composite outcome between the intervention and placebo groups containing the minimally-important clinical difference on a CNS Vital Signs composite measure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Laboratory-confirmed SARS-CoV-2 infection prior to randomization (we will track the specific date at which Covid-19 was diagnosed)
3. Presence of objective cognitive impairment (less than 18 on the MOCA-Blind) and/or the presence of subjective cognitive decline via the IQCODE-Short Form, as reflected in a score greater than 3.3.

Exclusion Criteria:

1. Non-English speaking
2. Incarcerated
3. Blind/ color blind
4. Unable to play the game due to a physical disability
5. Unable to play the game due to severe cognitive impairment (e.g., too inattentive or delirious) prior to randomization.
6. A known cognitive condition such as progressive dementia that would likely prevent the participant from responding to the effects of cognitive training or prevent them from being able to engage in self-consent.
7. Previously enrolled in a study using AKL-T01
8. Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable trial patient or unlikely to complete the trial.
9. Any other clinical condition that would jeopardize patient's safety while participating in this trial or may prevent the patient from adhering to the trial protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Improve cognition | 4 weeks
  To evaluate the feasibility of conducting a randomized trial evaluating the effectiveness of a digital app-based intervention (AKL-T01) to improve 4-week cognition (post-intervention) in cognitively impaired survivors of Covid-19.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided